CLINICAL TRIAL: NCT01422044
Title: Risk Prediction in Aortic Stenosis by Cardiac Autonomic Function
Brief Title: Risk Prediction in Aortic Stenosis
Acronym: PREDICT-AS
Status: Completed | Type: Observational
Sponsor: Thebiosignals.com (Other)
Responsible Party: Principal Investigator, Axel Bauer, Prof. Dr. med. Axel Bauer, Thebiosignals.com
Other Study IDs: 402/2009BO2-1
Record Dates: First submitted 2011-07-19; First posted 2011-08-23 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; autonomic function
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to test the prognostic value of autonomic markers in patients with aortic stenosis.

DETAILED DESCRIPTION:
Autonomic function will be assessed by presence of severe autonomic failure (defined by combination of abnormal heart rate turbulence and deceleration capacity).

Autonomic function will also be assessed by respiration and repolarization abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve area ≤1.5 qcm or mean aortic gradient ≥25mmHg

Exclusion Criteria:

* life expectancy <1 year due to non-cardiac causes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with at least moderate aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Total mortality | 2 years

SECONDARY OUTCOMES:
Cardiovascular mortality | 2 years
Combination of cardiovascular mortality and cardiac adverse events | 2 years
Correlation of presence of autonomic dysfunction with severity of aortic stenosis | at time of cardiac catheterization, which will be performed at an expected average of 3 days after hospital admission
  It will be assessed whether patients with cardiac autonomic dysfunction have more severe aortic stenosis.
  Autonomic dysfunction will assumed to be present when patients suffer from "severe autonomic failure" (i.e. combination of abnormal Heart Rate Turbulence and Deceleration Capacity).
  Severity of aortic stenosis will be assessed by clinical (symptoms, NYHA class), hemodynamic (mean aortic gradient, aortic valve area) and biochemical (Nt-BNP, high sensitive troponins) markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Klinik III, Tübingen, Germany

REFERENCES:
- [Derived] Zuern CS, Eick C, Rizas KD, Stoleriu C, Barthel P, Scherer C, Muller KA, Gawaz M, Bauer A. Severe autonomic failure in moderate to severe aortic stenosis: prevalence and association with hemodynamics and biomarkers. Clin Res Cardiol. 2012 Jul;101(7):565-72. doi: 10.1007/s00392-012-0427-3. Epub 2012 Feb 24. PMID 22362502